CLINICAL TRIAL: NCT01996670
Title: Early NCPAP Before Surfactant Treatment in Very Preterm Infants With RDS
Status: Completed | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Huiyi Huo, Department of Neonatology, Xiangya Hospital of Central South University
Other Study IDs: huohuiyi20131121; huo20131121 (Registry Identifier: huohuoyi)
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2007-01

CONDITIONS: Nasal Continuous Positive Airway Pressure,; Preterm Infants,; Surfactant Treatment,; Respiratory Distress Syndrome,; Bronchopulmonary Dysplasia
MeSH Terms: conditions — Respiratory Distress Syndrome; Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- <2h group
- 2-4h group
- >4h group

SUMMARY:
We hypothesis a period of early NCPAP before surfactant treatment is effective for treating RDS and preventing BPD in very premature infants.

ELIGIBILITY:
Inclusion Criteria:

* All enrolled infants were able to breathe at 5 min of age, had evidence of respiratory distress, unable to receive surfactant therapy, and were administrated with early NCPAP as the initial treatment

Exclusion Criteria:

* Exclusion criteria were endotracheal intubation for resuscitation or insufficient respiratory drive, died in the first 24 hours after birth, known genetic disorders, potentially life-threatening conditions unrelated to prematurity, and premature rupture of membranes (PROM) for >3 weeks.

Ages: 30 Minutes to 2 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: inborn infants at 26-32 weeks gestation with RDS, whom received NCPAP as the initial treatment, followed by surfactant treatment within 24 h after birth
Sampling Method: Non-Probability Sample
Enrollment: 683 (Actual)
Dates: Start 2007-01; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
death or bronchopulmonary dysplasia | 24 hours after birth